CLINICAL TRIAL: NCT03572686
Title: Comparison of the Effects of Adding Dexamethasone at 0.25% Ropivacaine With 0.5% Ropivacaine Alone in the Supraclavicular Brachial Plexus Block
Brief Title: Dexamethasone at Lower Concentration Ropivacaine in the Supraclavicular Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KMUHIRB-F(I)-20180034
Record Dates: First submitted 2018-06-03; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-04

CONDITIONS: Analgesia; Motor Activity; Brachial Plexus Block
Keywords: supraclavicular nerve block; dexamethasone; Ropivacaine
MeSH Terms: conditions — Agnosia; Motor Activity | interventions — Ropivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Ropivacaine High (RH) (Sham Comparator): Ultrasound-guided supraclavicular brachial plexus block with Ropivacaine 0.5% 20ml + N/S 1.6mL.
  Interventions: Drug: Ropivacaine 0.5% 20mL
- Group Ropivacaine Low (RL) (Placebo Comparator): Ultrasound-guided supraclavicular brachial plexus block with Ropivacaine 0.25% 20ml + N/S 1.6mL.
  Interventions: Drug: Ropivacaine 0.25% 20ml
- Group Ropivacaine Low + Dexamethasone (RLD) (Experimental): Ultrasound-guided supraclavicular brachial plexus block with Ropivacaine 0.25% 20ml + Dexamethasone 8mg (1.6mL).
  Interventions: Drug: Ropivacaine 0.25% 20ml + dexamethasone 8mg

INTERVENTIONS:
Drug: Ropivacaine 0.5% 20mL — In Group RH, participants received supraclavicular brachial plexus block with ropivacaine 0.5% 20ml at the end of surgery.
  Other Names: Ropivacaine high concentration 20ml
  Arms: Group Ropivacaine High (RH)
Drug: Ropivacaine 0.25% 20ml — In Group RL, participants received supraclavicular brachial plexus block with ropivacaine 0.25% 20ml at the end of surgery.
  Other Names: Ropivacaine low concentration 20ml
  Arms: Group Ropivacaine Low (RL)
Drug: Ropivacaine 0.25% 20ml + dexamethasone 8mg — In Group RLD, participants received supraclavicular brachial plexus block with ropivacaine 0.25% 20ml + dexamethasone 8mg at the end of surgery.
  Other Names: Ropivacaine low concentration 20ml + dexamethasone 8mg
  Arms: Group Ropivacaine Low + Dexamethasone (RLD)

SUMMARY:
The supraclavicular brachial plexus block is widely used in upper limb surgery below the shoulder. However, this can easily lead to long-term motor nerve blockage, Horner's syndrome, phrenic nerve paralysis or systemic poisoning, and even serious side effects such as cardiac arrest.

Dexamethasone is a synthetic corticosteroid and becoming more common to use steroids as an adjunct to local anesthetics in brachial plexus block.

In order to reduce the incidence of long-acting topical anesthetics from the nerve block in the supraclavicular arm, reducing the local anesthetic concentration is a feasible method, but this will also result in a shorter time to neurological block. The investigators hypothesized that the addition of Dexamethasone 5 mg to low concentrations (0.25%) of Ropivacaine would prolong postoperative analgesia.Therefore, the purpose of this study was to compare the postoperative analgesia and the side effects of postoperative supraclavicular brachial plexus blockade with the addition of Dexamethasone 5mg to Ropivacaine (0.5%) alone and Ropivacaine (0.25%) in low concentrations.

DETAILED DESCRIPTION:
The supraclavicular brachial plexus block is widely used in upper limb surgery below the shoulder. Although it is easier and more stable than axillary nerve block and subclavian brachial plexus block, long-acting local anesthetics are used for long-term blockade with traditional block methods. However, this can easily lead to long-term motor nerve blockage, Horner's syndrome, phrenic nerve paralysis or systemic poisoning, and even serious side effects such as cardiac arrest.

Ropivacaine is a novel long-acting topical amine amine topical anesthetics that lasts long and has anesthetic and analgesic effects. Its pharmacological characteristics are low cardiotoxicity, sensory block and motor block separation at low concentrations more obvious, and with the external peripheral vasoconstriction. Therefore, the drug is especially suitable for postoperative analgesia. Dexamethasone is a synthetic corticosteroid for the treatment of a wide range of symptoms including rheumatic diseases, certain skin diseases, severe allergies, asthma, chronic obstructive pulmonary disease, cerebral edema, and may also be combined with antibiotics for tuberculosis patients. It is becoming more common to use steroids as an adjunct to local anesthetics in brachial plexus block. Steroids have neurological blockade effects by blocking the nociceptive transmission of pith-type C-fibers and inhibiting the release of ectopic neurons. Dexamethasone, as a local anesthetic adjuvant in peripheral nerve block, has also been widely studied recently.

In order to reduce the incidence of long-acting topical anesthetics from the nerve block in the supraclavicular arm, reducing the local anesthetic concentration is a feasible method, but this will also result in a shorter time to neurological block. The investigators hypothesized that the addition of Dexamethasone 5 mg to low concentrations (0.25%) of Ropivacaine would prolong postoperative analgesia. Therefore, the purpose of this study was to compare the postoperative analgesia and the side effects of postoperative supraclavicular brachial plexus blockade with the addition of Dexamethasone 5mg to Ropivacaine (0.5%) alone and Ropivacaine (0.25%) in low concentrations.

ELIGIBILITY:
Inclusion Criteria:

* American society of Anesthesiology classification: I ~ III
* patients who have undergone arm surgery for blockage of the upper clavicle from nerve block

Exclusion Criteria:

* Patients had brachial plexus degeneration, coagulation abnormalities, obvious heart, lung, liver or kidney disease, body mass index less than 18.5 or greater than 35, body weight greater than 80 kg, pregnancy, regular use of steroids or opiates Opioids, chronic medication or alcohol abuse, as well as previous allergies or adverse reactions to opiates, dexamethasone, or the use of topical anesthetic Ropivacaine, were excluded from this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-04-13 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
analgesic effects (the intensity of pain) | 24 hours after the end of surgery
  The intensity of pain was assessed using a 0 to 10 Numerical Rating Scale (NRS) to quantify their degree of pain; where 0 means no pain and 10 conceivably the worst pain.

SECONDARY OUTCOMES:
blood pressure | 1 hour after the end of surgery
  systolic, diastolic, and mean blood pressure in the recovery room
motor block | 24 hours after the end of surgery
  Motor nerve block is evaluated using Lovett Rating Scale. 0 = complete blockage, 1 = almost complete blockage, 2 = significant motion impairment, 3 = mild motion impairment, 4 = significant loss of strength, 5 = slight decrease in strength, 6 = normal strength.
heart rate | 1 hour after the end of surgery
  heart rate in the recovery room

OTHER OUTCOMES:
postoperative nausea | 24 hours after the end of surgery
  Nausea was graded as 0 = none, 1 = mild, 2 = moderate, and 3 = severe.
postoperative vomiting | 24 hours after the end of surgery
  vomiting was graded as 0 = no, 1 = 1, 2 = 2, and 3 = 3 or more episodes

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Te Hsu, MD/PhD, Study Director — Department of anesthesiology,Kaohsiung Municipal Ta-Tung Hospital , Kaohsiung City 801，Taiwan (R.O.C.)
Locations (2):
- Taiwan (2):
  - Kaohsiung Municipal Ta-Tung Hospital, Kaohsiung City
  - Kaohsiung Medical University Hosptial, Kaohsiung City

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data.